CLINICAL TRIAL: NCT03052712
Title: Validation and Standardization of a Battery Evaluation of the Socio-emotional Functions in Various Neurological Pathologies
Acronym: GREFEXII
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2015_843_0031
Record Dates: First submitted 2017-02-07; First posted 2017-02-14 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer Disease; Parkinson Disease; Frontal Dementia; Huntington Disease; Traumatic Brain Injury; Stroke
Keywords: Disorders of socio-emotional; Alzheimer; frontal temporal dementia; Parkinson; Huntington; traumatic brain injury; stroke; focal lesions
MeSH Terms: conditions — Alzheimer Disease; Parkinson Disease; Huntington Disease; Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Active Comparator): battery of tests of social cognition
  Interventions: Behavioral: social cognition
- Control (Active Comparator): battery of tests of social cognition
  Interventions: Behavioral: social cognition

INTERVENTIONS:
Behavioral: social cognition — battery of tests of social cognition

SUMMARY:
The role of disorders of socio-emotional processes in cerebral diseases such as Alzheimer's disease, frontal temporal dementia, Parkinson's disease, Huntington's disease, traumatic brain injury, stroke, focal lesions, has been recognized recently. Social cognition refers to a large group of emotional and cognitive abilities regulating inter-individuals relationships and it includes mainly theory of mind, emotional information processing and empathy. However, assessment of socio-emotional processes is still largely based on experimental tests that are not validated for clinical purpose. In addition their long duration of administration is not adapted to clinical examination. Finally these tests have not been standardized and normalized in French-speaking population.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF)
2. Male or female, aged 20 to 80 years inclusive at the time of signing ICF
3. French-speaking
4. reliable informant

   Controls:
5. derived from the general population and consenting to participate in the study

   Patients:
6. MMS>18
7. Patients followed for mild or major neurocognitive disorder related to :

   * Alzheimer's disease
   * Frontotemporal lobar degeneration
   * Lewy bodies disease
   * Parkinson's disease
   * Huntington's disease
   * Progressive supranuclear palsy
   * traumatic brain injury
   * stroke or cerebral anoxia
   * mixed diseases
   * focal cerebral diseases

Exclusion Criteria:

1. Illiteracy
2. mental retardation
3. visual or motor deficit preventing reading, drawing or writing (scores on the reading, drawing or sentence writing subtests of the MMSE = 0)
4. hearing impairment interfering with understanding of instructions,
5. history of brain disease, including head injury with loss of consciousness lasting > 15 minutes, stroke, coma or loss of consciousness lasting > 15 minutes, followed for sclerosis or other brain disease, brain radiation therapy, epilepsy currently requiring treatment
6. history of psychiatric illness (schizophrenia or other psychosis) or ongoing psychiatric illness (major depressive disorder or other condition) currently requiring treatment or requiring a stay > 2 days in a psychiatry unit or anxiety requiring more than one medication at the present time
7. alcoholism (mean alcohol consumption > 3 standard drinks/day or history of alcohol withdrawal)
8. use of opiates or other illicit drugs during the previous 3 months or causing withdrawal syndrome
9. ongoing antidepressant or antiepileptic treatment
10. anxiolytic or hypnotic treatment initiated or increased during the previous month
11. general anaesthesia during the previous 3 months
12. history of heart surgery with cardiopulmonary bypass
13. comorbidities affecting cognition (respiratory, renal, liver, heart failure…)
14. women of childbearing potential (defined as pre-menopausal, less than 2 years postmenopausal, or not surgically sterile)
15. persons placed under judicial protection

    Patients :
16. contraindication to MRI

    Controls:
17. deficit on MMSE <27

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2016-09-09 (Actual); Primary Completion 2019-09-08 (Actual); Study Completion 2019-09-08 (Actual)

PRIMARY OUTCOMES:
tests of social cognition (questionnaire) | 3 years
  standardize and validate in French-speaking population a comprehensive battery of tests of social cognition

CONTACTS AND LOCATIONS:
Overall Officials: Olivier GODEFROY, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France